CLINICAL TRIAL: NCT01807156
Title: Phase II Trial of Tivozanib in Advanced Hepatocellular Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Primary endpoint not met
Sponsor: Emory University (Other)
Collaborators: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Bassel El-Rayes, Study Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00061422; IRB00061422 (Other: Emory University); WINSHIP2302-12 (Other: Other)
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Results first posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Cancer
Keywords: Tivozanib; Advanced hepatocellular cancer; Angiogenesis
MeSH Terms: conditions — Liver Neoplasms | interventions — tivozanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tivozanib (Experimental): Patients would receive Tivozanib 1.0 mg/day orally, 3 weeks on, one week off, for one cycle starting day 1. If no adverse event is encountered, patients will continue subsequent cycles of Tivozanib 1.5 mg/day orally; 3 weeks on/1 week off, dosing schedule. Patients will continue on treatment until disease progression, unacceptable toxicity, or patient withdrawal from the study.
  Interventions: Drug: Tivozanib

INTERVENTIONS:
Drug: Tivozanib — Oral medication given daily. No placebo.
  Other Names: AV-951

SUMMARY:
The purpose of this study is to learn about the effect of the investigational agent tivozanib on the control of the tumor growth in hepatocellular (liver) cancer. The investigators also plan to collect information on the likelihood to develop side effects while on this treatment. Tivozanib is an oral medication (pill) taken once a day. This medication is designed to stop the tumor from developing new blood vessels.

DETAILED DESCRIPTION:
Angiogenesis is the formation of new blood vessels. Angiogenesis is driven by cytokines including vascular endothelial growth factor. Tivozanib is an oral medication that inhibits vascular endothelial growth factor preventing tumor from developing new blood vessels.

The purpose of this study is to evaluate the effects of tivozanib on hepatocellular (liver) cancer. Participants in the study take tivozanib daily at a dose of 1 mg for 1month. if doing well the dose would be increased to 1.5 mg per day. Patients are monitored for response using CT or MRI scans every 2months. In addition, patients will have blood draws to evaluate the effects of tivozanib on blood vessels.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with measurable, histological diagnosis of hepatocellular carcinoma (HCC) and whose disease is not amenable to surgical or regional therapy.
2. Prior allowed therapy:

   * Surgery including hepatic resection

     1. Minimum of 4 weeks since any surgical procedure.
     2. Patients must have adequately recovered from surgery.
   * Regional therapy

     1. Includes transarterial chemoembolization (TACE), drug-eluting bead [DEB]-TACE, percutaneous ethanol injection, radiofrequency/cryo ablation, Yttrium-90 radioembolization.
     2. More than 2 weeks must have lapsed from therapy.
     3. There must be an indicator lesion outside the treated area or clear evidence of progression in the treated lesion, not amenable for further local therapies.
     4. Concomitant sorafenib with regional therapy is allowed as long as no evidence of progression on sorafenib.
   * Prior adjuvant sorafenib is allowed, if completed more than 6 months prior to disease recurrence.
3. Adequate hematological, liver and metabolic organ function.
4. Signed informed consent.

Exclusion Criteria:

1. Patients with mixed histology or fibrolamellar variant.
2. Prior systemic therapy for metastatic disease.
3. Uncontrolled hypertension (HTN).
4. Symptomatic heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bassel El-Rayes, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University, Winship Cancer Institute, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tivozanib
Started | 7
Completed | 6
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tivozanib
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: years] | 55 [31 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Advanced Hepatocellular Cancer (HCC) Receiving Tivozanib Who Are Free From Progression
Description: Evaluation of disease progression in the patients with advanced hepatocellular cancer (HCC) receiving tivozanib will be made using CT or MRI scan of the organ(s) with the target lesion(s). Response Evaluation Criteria In Solid Tumors (RECIST) criteria 1.1 will be used for objective tumor response assessment. Measurable lesions can be measured in at least one dimension as ≥ 20 mm with conventional CT scan techniques or as ≥ 10 mm with spiral CT scan. Target lesions are all measurable lesions up to a maximum of 5 lesions. Target lesions are selected for their size and suitability for accurate repetitive measurements. The sum of the longest diameter of all target lesions will be calculated and reported as the baseline sum longest diameter (LD). This will be used as a reference to further quantify objective response.
Time Frame: 6 Months
Measure: Number; unit: participants
Arm/Group | Tivozanib
Number analyzed (Participants) | 6
participants | 1

2. Secondary Outcome: Response Rate Based on Response Evaluation Criteria in Solid Tumors (RECIST) Criteria
Description: Measurable lesions: Lesions that can be measured in at least one dimension as ≥ 20 mm with conventional CT scan techniques or as ≥ 10 mm with spiral CT scan.
  Non-measurable lesions: All other lesions including small lesions (longest diameter < 20 mm with conventional techniques) and other non-measurable lesions including: pleural effusions, ascites, and disease documented by indirect evidence (e.g. biochemical abnormalities).
  Target lesions: All measurable lesions up to a maximum of 5 lesions. Target lesions are selected for their size and suitability for accurate repetitive measurements. The sum of the longest diameter of all target lesions will be calculated and reported as the baseline sum longest diameter (LD). This will be used as a reference to further quantify objective response.
  Non-target lesions: All other lesions are identified as non-target lesions and should be followed as present or absent.
Time Frame: 6 months
Population: No response was observed in any of the patients.
Measure: Number; unit: participants
Arm/Group | Tivozanib
Number analyzed (Participants) | 6
participants | 0

ADVERSE EVENTS:
Arm/Group | Tivozanib
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tivozanib (N=7)
Pulmonary Embolism (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tivozanib (N=7)
Liver Function Test Elevation (Hepatobiliary disorders) | 1
Hypertension (Cardiac disorders) | 3
Nausea (General disorders) | 1
Fatigue (General disorders) | 1
Headache (Nervous system disorders) | 1
Insomnia (General disorders) | 2
Abdominal Pain (General disorders) | 1
Hyperglycemia (Blood and lymphatic system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes